CLINICAL TRIAL: NCT03359057
Title: Trial Evaluating Folic Acid Supplementation by Concomitant Administration of Ethinyl Estradiol + Levonorgestrel (Ethinyl Estradiol + Levonorgestrel + Folic Acid - Coated Tablet - 0.02 mg + 0.10 mg + 0.4 mg; Biolab Sanus Farmaceutica Ltda) in Female Volunteers.
Brief Title: Trial Evaluating Folic Acid Supplementation by Concomitant Administration of Ethinyl Estradiol + Levonorgestrel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galeno Desenvolvimento de Pesquisas Clínicas (Other Government)
Collaborators: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Principal Investigator, Gilberto De Nucci, Doctor, Galeno Desenvolvimento de Pesquisas Clínicas
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDN 028/12
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Contraception
Keywords: Folic acid; Supplementation; Ethinyl estradiol; Levonorgestrel; Oral contraceptive
MeSH Terms: interventions — Ethinyl Estradiol; Levonorgestrel; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estradiol + levonorgestrel + folic acid (Experimental): Coated tablet of the test product - ethinyl estradiol + levonorgestrel + folic acid, 0.02 mg + 0.10 mg + 0.4 mg for 21 days.
  Interventions: Drug: ethinyl estradiol + levonorgestrel + folic acid
- Folic acid (Placebo Comparator): Coated tablet of placebo coated tablet containing folic acid 0.4 mg only on the last 7 days of the cycle.
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: ethinyl estradiol + levonorgestrel + folic acid — One coated tablet of ethinyl estradiol + levonorgestrel + folic acid, 0.02 mg + 0.10 mg + 0.4 mg for 21 days in 3 cycles (12 weeks).
  Arms: Estradiol + levonorgestrel + folic acid
Drug: Folic Acid — One coated tablet of folic acid 0.4 mg for 7 days in 3 cycles (12 weeks).
  Arms: Folic acid

SUMMARY:
This trial evaluated folic acid supplementation after oral administration of the ethinyl estradiol + levonorgestrel + folic acid (0.02 mg + 0.10 mg + 0.4 mg) coated tablet (Level-Fol® Biolab Sanus Farmacêutica, São Paulo, Brazil) in healthy female volunteers, based on statistical comparisons of folate levels in erythrocytes. Its safety and tolerability was also evaluated.

DETAILED DESCRIPTION:
This Phase III trial was performed as a monocentric, open label, randomized design, with 1 treatment regimen, in 3 cycles (12 weeks), with administration in multiple doses, in which the healthy volunteers received one coated tablet of the test product - ethinyl estradiol + levonorgestrel + folic acid, 0.02 mg + 0.10 mg + 0.4 mg (Level-Fol® Biolab Sanus Farmaceutica, Brazil) for 21 days and a placebo coated tablet containing folic acid 0.4 mg only (Biolab Sanus Farmaceutica, Brazil) on the last 7 days of the cycle.

The subjects were required to present to the Clinical Unit for every drug administration, which was assisted by a member of the research team. Blood samples of 15 mL were collected via direct venepuncture into tubes containing 50 µL of ethylenediaminetetraacetic acid (EDTA) at pre-dose, 1st, 21st, 28th, 29th, 49th, 56th, 57th, 77th and 84th day of treatment.

Te safety assessment was based on recording adverse events throughout the study duration as well as through the monitoring of vital signs and evaluation of laboratory tests and ECG.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers aged between 18 and 35 years old (fertile age), without hormonal contraceptive use at least 3 months (oral) or 1 year (injectable), regular cycle and no pregnant or breastfeeding;
* Body mass index (BMI) ≥ 19.0 kg/m² and ≤ 28.75 kg/m²
* No evidence of significant diseases, that, at the investigator's discretion, may affect the participation in the clinical trial, in accordance with the protocol requirements
* Ability to understand the nature and the objective of the clinical trial, including the risks and possible side effects; intention to cooperate with the investigator and act in accordance with the protocol requirements, as confirmed by the informed consent form signature.

Exclusion Criteria:

* Subjects with known hypersensitivity to the compounds of the investigational products, severe allergies or multiple drug allergies
* Existing diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the drug
* Screening laboratory tests presenting deviations deemed as clinically significant, which, due to possible risks, prevents the participation in clinical trial.
* Use of maintenance therapy with any drug
* Drug or alcohol dependence
* Volunteers who ingests more than 5 cups of coffee or tea per day and/or smoke
* Volunteers with unusual eating habits, e.g, vegetarian
* Treatment, within 3 months prior to the initiation of the clinical trial treatment, with any drug known to have a well-established toxic potential to major organs.
* Use of regular medication within 2 weeks before the start of treatment and the date of evaluation, or made use of any medication within one week, except for oral contraceptives or cases where, based on the half-life of the drug and/or active metabolites, complete elimination can be assumed
* Treatment within 6 months prior to the study with any known drug of have a well-defined toxic potential in large organs
* Hospitalization for any reason up to 8 weeks before the start of the treatment of this study
* Participation in a clinical trial during the last 6 months
* Blood donation or other blood loss of more than 450 mL within the last 3 months
* Pregnant, delivery or abortion in the 12 weeks prior to the planned hospitalization
* The volunteer who has any condition that prevents him from participating in the study by judgment of the investigator

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-02-26 (Actual); Primary Completion 2013-07-04 (Actual); Study Completion 2013-09-17 (Actual)

PRIMARY OUTCOMES:
Measurement of folate levels in erythrocytes. | 0-84 days
  Blood sampling for the determination of erythrocyte levels of folate in the subjects after the treatment with the test drug or placebo.

SECONDARY OUTCOMES:
Number of adverse events | 0-84 days
  Number of adverse events, including clinically relevant alterations of vital signs and laboratory tests results

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, Doctor, Principal Investigator — Galeno Desenvolvimento de Pesquisas Clinicas Ltda
Locations (1):
- Galeno Desenvolvimento de Pesquisas Clinicas Ltda. - ME, Campinas, São Paulo, Brazil